CLINICAL TRIAL: NCT06390111
Title: A Phase 4, Multi-center, Open Label Trial to Evaluate Efficacy of Reinduction With Nadofaragene Firadenovec in Subjects With CIS ± High-grade Ta/T1 and no Complete Response to First Nadofaragene Firadenovec Dose.
Brief Title: A Trial to Evaluate Efficacy of Reinduction With Nadofaragene Firadenovec in Subjects With CIS ± High-grade Ta/T1 and no Complete Response to First Nadofaragene Firadenovec Dose.
Acronym: ABLE-42
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Ferring decided to prioritize collection of ADSTILADRIN re-induction data in patients with HR BCG-unresponsive NMIBC who did not have a CR to the initial dose of ADSTILADRIN through data sources within the clinical setting including ABLE-22 and -41.
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 000439
Record Dates: First submitted 2024-04-19; First posted 2024-04-30 (Actual); Last update posted 2024-11-22 (Actual); Status verified 2024-08

CONDITIONS: Bladder Cancer; Ta/T1; CIS
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nadofaragene Firadenovec (Experimental): Eligible subjects will receive nadofaragene firadenovec. This will be instilled quarterly in the bladder followed by quarterly disease assessments.
  Interventions: Drug: nadofaragene firadenovec

INTERVENTIONS:
Drug: nadofaragene firadenovec — The investigational medicinal product dose, concentration, and assessments are aligned with nadofaragene firadenovec US prescribing information.
  Other Names: Adstiladrin

SUMMARY:
In this phase 4 trial (000439), subjects with NMIBC CIS (± high-grade Ta/T1) who have not responded to their first dose of nadofaragene firadenovec (commercial ADSTILADRIN received before trial entry) will be offered reinduction when entering the trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed, as documented, with CIS ± high-grade disease Ta/T1 and absence of progression after first dose of nadofaragene firadenovec within the last 5 months from instillation.
* Diagnosed, as documented, with:

  * Low risk of disease progression as assessed at the discretion of the investigator
  * Previous Bacillus Calmette Guerin (BCG) therapy (BCG exposed) with no maximum limit to the amount of BCG administered

Exclusion Criteria:

* Current or previous evidence of muscle-invasive (muscularis propria) or metastatic disease presented at the screening visit. Examples of increased risk of muscle-invasive include but are not limited to:

  * Presence of lymphovascular invasion and / or micropapillary disease as shown in the histology of the biopsy sample
  * Subjects with T1 disease accompanied by the presence of hydronephrosis secondary to the primary tumor
* Current and prior systemic or local therapy for bladder cancer since first dose of nadofaragene firadenovec
* Current or prior investigational treatment for BCG-unresponsive NMIBC or any other investigational drug (drug used in a clinical trial, i.e drug used in a Ferring sponsored non-interventional study does not apply) since first dose of nadofaragene firadenovec
* Clinically significant and unexplained elevated liver or renal function tests
* History of malignancy of other organ system within past 5 years, except treated basal cell carcinoma or squamous cell carcinoma of the skin and ≤pT2 upper tract urothelial carcinoma at least 24 months after nephroureterectomy. Also subjects with genitourinary cancers other than urothelial cancer or prostate cancer that are under active surveillance are excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Complete response (CR) achieved at month 3 after nadofaragene firadenovec retreatment | at month 3

SECONDARY OUTCOMES:
Maintenance of CR at months 6 after nadofaragene firadenovec retreatment | at 6 months after nadofaragene firadenovec retreatment
Maintenance of CR at months 9 after nadofaragene firadenovec retreatment | at 9 months after nadofaragene firadenovec retreatment
Maintenance of CR at months 12 after nadofaragene firadenovec retreatment | at 12 months after nadofaragene firadenovec retreatment
Durability of CR at months 6 after nadofaragene firadenovec retreatment | at 6 months after nadofaragene firadenovec retreatment
  No evidence of CIS and/or high-grade Ta/T1
Durability of CR at months 9 after nadofaragene firadenovec retreatment | at 9 months after nadofaragene firadenovec retreatment
  No evidence of CIS and/or high-grade Ta/T1
Durability of CR at months 12 after nadofaragene firadenovec retreatment | at 12 months after nadofaragene firadenovec retreatment
  No evidence of CIS and/or high-grade Ta/T1
Muscle-invasive progression of disease up to month 12 after nadofaragene firadenovec retreatment | Up to12 months after nadofaragene firadenovec retreatment
Incidence of cystectomy | Up to 12 months after nadofaragene firadenovec retreatment
Time to cystectomy | Up to 12 months after nadofaragene firadenovec retreatment
Pathological staging at cystectomy | Up to 12 months after nadofaragene firadenovec retreatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (2):
- United States (2):
  - Ferring Investigational Site, Little Rock, Arkansas
  - Ferring Investigational Site, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No